CLINICAL TRIAL: NCT00099242
Title: Efficacy and Safety of the Rivastigmine Transdermal Patch in Patients With Probable Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CENA713D2320
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Alzheimer's Disease; Dementia, Alzheimer Type
Keywords: Alzheimer's Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

INTERVENTIONS:
Drug: rivastigmine transdermal patch

SUMMARY:
The goal of this research study is to evaluate the safety and efficacy of the rivastigmine transdermal patch in patients with probable Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia of the Alzheimer's type
* Males, and females who are surgically sterile or one year postmenopausal
* A primary caregiver willing to accept responsibility for supervising the treatment

Exclusion Criteria:

* Any condition (other than Alzheimer's) that could explain patient's dementia
* An advanced, severe or unstable disease that may put the patient at special risk
* Current diagnosis of active, uncontrolled seizure disorder or unstable cardiovascular disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040
Dates: Start 2003-11; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Change in cognition from baseline at week 24
Global clinical impression of change from baseline at week 24

SECONDARY OUTCOMES:
Change from baseline at week 24 in activities of daily living
Change from baseline at week 24 in behavioral symptoms
Change from baseline at week 24 in global cognitive testing
Change from baseline at week 24 in executive function
Change from baseline at week 24 in attention

CONTACTS AND LOCATIONS:
Locations (75):
- United States (22):
  - Orange, California
  - San Francisco, California
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Port Charlotte, Florida
  - West Palm Beach, Florida
  - Snellville, Georgia
  - St Louis, Missouri
  - Omaha, Nebraska
  - Long Branch, New Jersey
  - Toms River, New Jersey
  - Whiting, New Jersey
  - Columbus, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Greensburg, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Tacoma, Washington
- Chile (2):
  - Santiago
  - Valparaíso
- Czechia (5):
  - Brno
  - Brno-Bohunice
  - Hradec Králové
  - Olomouc
  - Prague
- Denmark (3):
  - Copenhagen
  - Glostrup Municipality
  - Hillerød
- Kuopio, Finland
- Investigative Sites, Germany
- Guatemala City, Guatemala
- Israel (5):
  - Beersheva
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
- Italy (3):
  - Lido di Camaiore
  - Milan
  - Pescara
- Mexico (3):
  - Guadalajara Jalisco
  - Mexico City
  - Monterrey Nuevo Leon
- Norway (4):
  - Bodø
  - Oslo
  - Tromsø
  - Trondheim
- Lima, Peru
- Poland (5):
  - Gdansk
  - Lublin
  - Poznan
  - Szczecin
  - Warsaw
- Portugal (2):
  - Amadora
  - Coimbra
- Bayamón, Puerto Rico
- Russia (2):
  - Moscow
  - Saint Petersburg
- Slovakia (2):
  - Bratislava
  - Michalovce
- South Korea (3):
  - Jungbuk
  - KyungKi-province
  - Seoul
- Sweden (4):
  - Gothenburg
  - Kalmar
  - Stockholm
  - Uppsala
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
- Ciudad Merida, Mérida, Venezuela

REFERENCES:
- [Derived] Lefevre G, Callegari F, Gsteiger S, Xiong Y. Effects of Renal Impairment on Steady-State Plasma Concentrations of Rivastigmine: A Population Pharmacokinetic Analysis of Capsule and Patch Formulations in Patients with Alzheimer's Disease. Drugs Aging. 2016 Oct;33(10):725-736. doi: 10.1007/s40266-016-0405-y. PMID 27681702
- [Derived] Alva G, Grossberg GT, Schmitt FA, Meng X, Olin JT. Efficacy of rivastigmine transdermal patch on activities of daily living: item responder analyses. Int J Geriatr Psychiatry. 2011 Apr;26(4):356-63. doi: 10.1002/gps.2534. PMID 21312297